CLINICAL TRIAL: NCT02078843
Title: Diagnostic Accuracy of Gallium-68-DOTATATE PET/CT Compared to Indium-111-pentetreotide Scintigraphy (SPECT/CT) for Gastroenteropancreatic Neuroendocrine Tumors
Acronym: GaIN
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Superiority of one imaging method
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: University of Lausanne Hospitals (Other); University Hospital, Basel, Switzerland (Other); University of Bern (Other); SWAN Isotopen AG, Bern (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 092/11
Record Dates: First submitted 2014-02-26; First posted 2014-03-05 (Estimated); Last update posted 2016-09-07 (Estimated); Status verified 2016-09

CONDITIONS: Gastroenteropancreatic Neuroendocrine Tumors
Keywords: NET; Gallium-68-DOTATATE; PET/CT; Indium-111-pentetreotide scintigraphy; octreoscan; GEP-NET; gastroenteropancreatic neuroendocrine tumors
MeSH Terms: conditions — Gastro-enteropancreatic neuroendocrine tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- All patients (Other): Subsequent performance of index test and standard test
  Interventions: Drug: Gallium-68-DOTATATE PET/CT (index test); Drug: Indium-111-Octreoscan (standard test)

INTERVENTIONS:
Drug: Gallium-68-DOTATATE PET/CT (index test) — Somatostatin-based imaging tracer
Drug: Indium-111-Octreoscan (standard test) — Somatostatin-based imaging tracer

SUMMARY:
The investigators hypothesize that the new imaging method Gallium-68-DOTATATE has a higher diagnostic value in the detection of neuroendocrine tumors than the established imaging method Indium-111-Octreoscan. Therefore, the investigators will perform both imaging procedures in patients with suspected or confirmed neuroendocrine tumors. Subsequently, the investigators will compare the diagnostic performance of both methods.

DETAILED DESCRIPTION:
Background

Neuroendocrine tumors Neuroendocrine tumors (NET) are heterogeneous slow-growing neoplasms, occurring in 1-4/100,000 people per year. They origin from endocrine cells that derive from entodermal stem cells and are characterized by an endocrine metabolism and a typical pathologic pattern.

Slow metabolic rates of NET, small lesion size and variable anatomical localization have represented the major limits for lesions diagnosis. The diagnostic workup for NET has relied on conventional morphological imaging procedures including computed tomography (CT), ultrasound (US) and magnetic resonance imaging (MRI) combined with gamma camera functional imaging, namely whole-body somatostatin receptor scintigraphy (SRS). SRS show a higher diagnostic accuracy than CT for NET diagnosis at both the primary and metastatic site, but there is still room for improvement. Novel PET tracers specifically developed for NET may increase diagnostic accuracy considerably as outlined below.

Somatostatin receptor scintigraphy (SRS) As NET have high affinity somatostatin receptors, scintigraphic methods have been developed in the early nineties to allow in vivo imaging. SRS using Indium-111-DTPA-octreotide (Indium-111-pentetreotide scintigraphy), is the most widely used diagnostic test. Although rather sensitive and helpful for whole body staging compared to traditional imaging methods, this technique has pitfalls, one of them being the poor spatial resolution, leading to the development of PET-based imaging.

Gallium-68-DOTA-peptide PET In the past decade, several positron emitting tracers have been developed for NET imaging. 68Ga-DOTA-peptides are a group of PET tracers that specifically bind to somatostatin receptors (SSTR) over-expressed on NET cells. Gallium-68-DOTA-peptides structure can be summarized in (1) the active part binding to SSTR (TOC, NOC, TATE), (2) the chelant (DOTA) and (3) the isotope (68Ga). Indications to perform 68Ga -DOTA-peptides studies in NET patients include: staging, re-staging after therapy, identification of the site of the unknown primary tumor in patients with proven NET secondary lesions and selection of cases eligible for therapy with somatostatin analogues.

68Ga-DOTA-TOC was the first tracer to be employed in NET imaging and was reported to present a high tumor to non-tumor contrast and a higher sensitivity compared to SRS . The study with the largest patients population (84 pts with NET), reported sensitivity (97%) for DOTA-TOC PET to be superior to CT (61%) and SRS (52%) for the detection of NET lesions, especially in case of small tumors at nodal or bone level. In a comparison study of 51 patients with well differentiated NET, PET with Gallium-DOTA-TOC performed better than CT and SRS for the early detection of bone NET secondary lesions (sensitivity of 97%, specificity of 92%). 68Ga-DOTA-TATE is characterized by a very high affinity for SSTR2 with a considerably higher affinity than 111In-DTPA octreotide. In a recent study, 51 patients with established NET (35 negative and 16 equivocal for uptake on SRS) were examined by 68Ga-DOTA-TATE PET. 68Ga-DOTA-TATE PET identified significantly more lesions than SRS and changed management in 36 patients (70.6%), who were subsequently deemed suitable for peptide receptor-targeted therapy.

Rationale of the study 111In-pentetreotide scintigraphy is the current standard for the detection of NET, even though its diagnostic accuracy is less than optimal. In the past decade, several 68Ga-DOTA-peptides have been developed for NET imaging, which showed a better detection for NET than 111In-pentetreotide scintigraphy in a small number of studies. These studies had several limitations, most importantly the inclusion of rather small and heterogeneous patient populations.

The aim of this study is to prospectively compare the diagnostic accuracy of 68Ga-DOTA-TATE PET/CT with 111In-pentetreotide scintigraphy in a well-defined population of consecutive patients with established GEP-NET or patients with suspicion of NET with indication for a scintigraphy.

Objective

The objective of this study is to compare the diagnostic accuracy of Gallium-68-DOTATATE PET/CT with Indium-111-pentetreotide scintigraphy (SPECT/CT) for the diagnosis of gastroenteropancreatic neuroendocrine tumors (GEP-NET) in consecutive patients with established GEP-NET or patients with suspicion of NET with indication for a scintigraphy. The working hypothesis is that Gallium-68-DOTATATE PET/CT is superior to Indium-111-pentetreotide scintigraphy (SPECT/CT) in terms of sensitivity and specificity.

Methods

The present study is a multi-center assessor-blind diagnostic case-control study of Gallium-68-DOTATATE PET/CT compared to Indium-111-pentetreotide scintigraphy (SPECT/CT) in consecutive patients with established GEP-NET or patients with suspicion of NET with indication for a scintigraphy.

The study is conducted at the University Hospital Basel, Bern University Hospital, and CHUV Lausanne. The University Clinics of Nuclear Medicine of Basel, Bern and Lausanne, as well as Endocrinology, Diabetes and Clinical Nutrition of Bern will accrue consecutive patients with established GEP-NET or patients with suspicion of GEP-NET that meet eligibility criteria. All patients will undergo Gallium-68-DOTATATE PET/CT as index test and Indium-111-pentetreotide scintigraphy as standard test. Both results will be compared with histology and the follow-up results as diagnostic gold standards.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Signed written informed consent with full understanding of the study procedures and the investigational nature of the study
* Patient referred to Indium-111-pentetreotide scintigraphy., which was performed as part of clinical routine care
* Inclusion criteria specific for cases only
* Histologically established GEP-NET (new or recurrent)
* Tumor mass remaining after initial biopsy or surgery
* Inclusion criteria specific for controls only
* 5.6. Suspicion of any NET (new or recurrent) but no established diagnosis or established diagnosis of any NET (new or recurrent) but no remaining tumor mass after surgery

Exclusion Criteria

* Previous inclusion in the same study with the following exception: a patient may be included as case if she/he was previously included as control
* Gastric type 2 ECL cell neuroendocrine tumors
* Pregnant or nursing women
* Known intolerance to any protocol required diagnostic intervention
* Patient's lack of accountability, inability to appreciate the nature, meaning and consequences of the study and to formulate his/her own wishes correspondingly
* Exclusion criteria specific for controls only
* Patients for whom it remains unclear whether the tumor was completely removed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2014-03; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Number of patients correctly identified as having GEP-NET by using Gallium-68-DOTATATE PET/CT and Indium-111-pentetreotide scintigraphy (SPECT/CT) | 6 months
Number of patients correctly identified as not having GEP-NET by using Gallium-68-DOTATATE PET/CT and Indium-111-pentetreotide scintigraphy (SPECT/CT) | 6 months

SECONDARY OUTCOMES:
Patient satisfaction | 6 months
  Measured by patient satisfaction questionnaire relating to Indium-111-pentetreotide scintigraphy
Number of patients with adverse events | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Krause, Prof. Dr. med., Principal Investigator — Institute of Nuclear Medicine, University Hospital Berne; Christoph Stettler, Prof. Dr. med., Principal Investigator — Division of Endocrinology, University Hospital Bern
Locations (1):
- Nuclear Medicine, Bern University Hospital, Bern, Switzerland

REFERENCES:
- [Background] Gabriel M, Oberauer A, Dobrozemsky G, Decristoforo C, Putzer D, Kendler D, Uprimny C, Kovacs P, Bale R, Virgolini IJ. 68Ga-DOTA-Tyr3-octreotide PET for assessing response to somatostatin-receptor-mediated radionuclide therapy. J Nucl Med. 2009 Sep;50(9):1427-34. doi: 10.2967/jnumed.108.053421. Epub 2009 Aug 18. PMID 19690033
- [Background] Putzer D, Gabriel M, Henninger B, Kendler D, Uprimny C, Dobrozemsky G, Decristoforo C, Bale RJ, Jaschke W, Virgolini IJ. Bone metastases in patients with neuroendocrine tumor: 68Ga-DOTA-Tyr3-octreotide PET in comparison to CT and bone scintigraphy. J Nucl Med. 2009 Aug;50(8):1214-21. doi: 10.2967/jnumed.108.060236. Epub 2009 Jul 17. PMID 19617343
- [Background] Antunes P, Ginj M, Zhang H, Waser B, Baum RP, Reubi JC, Maecke H. Are radiogallium-labelled DOTA-conjugated somatostatin analogues superior to those labelled with other radiometals? Eur J Nucl Med Mol Imaging. 2007 Jul;34(7):982-93. doi: 10.1007/s00259-006-0317-x. Epub 2007 Jan 16. PMID 17225119
- [Background] Reubi JC, Schar JC, Waser B, Wenger S, Heppeler A, Schmitt JS, Macke HR. Affinity profiles for human somatostatin receptor subtypes SST1-SST5 of somatostatin radiotracers selected for scintigraphic and radiotherapeutic use. Eur J Nucl Med. 2000 Mar;27(3):273-82. doi: 10.1007/s002590050034. PMID 10774879
- [Background] Srirajaskanthan R, Kayani I, Quigley AM, Soh J, Caplin ME, Bomanji J. The role of 68Ga-DOTATATE PET in patients with neuroendocrine tumors and negative or equivocal findings on 111In-DTPA-octreotide scintigraphy. J Nucl Med. 2010 Jun;51(6):875-82. doi: 10.2967/jnumed.109.066134. Epub 2010 May 19. PMID 20484441